CLINICAL TRIAL: NCT06665061
Title: Effects of Different Ventilation Modes on Airway Pressure and Intracranial Pressure in Patients in the Trendelenburg Position: a Randomized, Double-blind, Controlled Trial
Brief Title: Effects of Different Ventilation Modes on Airway Pressure and Intracranial Pressure in Patients in the Trendelenburg Position
Acronym: PCV、VCV、PRVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inner Mongolia Baogang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-MER-106; No. 2024MS08058 (Other Grant/Funding Number: Project of Natural Science Foundation of Inner Mongolia Autonomous Region); No. 2023wsjkkj120 (Other Grant/Funding Number: Baotou Health Research Project); No. YKD2024LH011 (Other Grant/Funding Number: Joint Project of Inner Mongolia Medical University)
Record Dates: First submitted 2024-10-13; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Laparoscopic Myomectomy
Keywords: Trendelenburg Position; pressure-controlled ventilation; volume-controlled ventilation; pressure-regulated volume-controlled ventilation; Optic nerve sheath diameter

STUDY DESIGN:
Intervention Model Description: This study enrolled patients aged 27-77 years who underwent elective laparoscopic myomectomy at our institution from February 2023 to August 2024. The patients had an ASA classification of I-III. Patients were excluded if they had an allergy to the anesthetic drugs used in the study, adverse effects to the analgesics included, liver cirrhosis or kidney dysfunction, or cardiopulmonary impairment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The anesthesiologists and surgeons performing the anesthesia and assisting with the surgery were only informed of the mechanical ventilation mode to be used. Patients were unaware of their group assignment because mechanical ventilation was initiated after anesthesia induction when they were unconscious. The anesthetic nurses and doctors evaluating the patients postoperatively were also unaware of the group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- PCV (Experimental): After intubation under anesthesia, mechanical ventilation is performed in the pressure control ventilation (PCV) mode.
  Interventions: Device: PCV
- VCV (Experimental): After intubation under anesthesia, mechanical ventilation is performed in the volume control ventilation (VCV) mode.
  Interventions: Device: VCV
- PRVC (Experimental): After intubation under anesthesia, mechanical ventilation is performed in the pressure-regulated volume control (PRVC) mode.
  Interventions: Device: PRVC

INTERVENTIONS:
Device: PCV — Patients were randomly assigned to receive PCV mechanical ventilation, with consistent ventilation parameters.
  Arms: PCV
Device: VCV — Patients were randomly assigned to receive VCV mode mechanical ventilation, with consistent ventilation parameters.
  Arms: VCV
Device: PRVC — Patients were randomly assigned to receive PRVC mode mechanical ventilation, with consistent ventilation parameters.
  Arms: PRVC

SUMMARY:
The goal of this clinical trial is to understand the impact of three different ventilation modes-pressure-controlled ventilation (PCV), volume-controlled ventilation (VCV), and pressure-regulated volume-controlled ventilation (PRVC)-on airway pressure and intracranial pressure in patients undergoing resuscitation positioning. It aims to evaluate the effects of these ventilation modes on patients in resuscitation positions. The main questions it seeks to answer are:

Does the PRVC mode more effectively control airway pressure and intracranial pressure in patients undergoing resuscitation positioning? Does it help to reduce the risk of increased intracranial pressure during surgery?

DETAILED DESCRIPTION:
2.1. Trial design This single-center, parallel-arm, double-blinded, randomized, noninferiority trial was performed at Inner Mongolia Baogang Hospital, The Third Affiliated Hospital of Inner Mongolia Medical University, China, from January 2022 to June 2024. The study adhered to Good Clinical Practice guidelines and the principles of the Declaration of Helsinki. 2.2. Participants This study enrolled patients aged 27-77 years who underwent elective laparoscopic myomectomy at our institution from February 2023 to August 2024. The patients had an ASA classification of I-III. Patients were excluded if they had an allergy to the anesthetic drugs used in the study, adverse effects to the analgesics included, liver cirrhosis or kidney dysfunction, or cardiopulmonary impairment. Patients were also excluded if they were uncooperative, defined as being unable to undergo clinical assessment. This study was approved by the Medical Ethics Committee of Inner Mongolia Baogang Hospital (2023-MER-106) .

2.3. Randomization and blinding Patients who met the inclusion criteria were randomly assigned to one of three groups (PCV, VCV, or PRVC) in a 1:1:1 ratio using a random number table. The anesthesiologists and surgeons performing the anesthesia and assisting with the surgery were only informed of the mechanical ventilation mode to be used. Patients were unaware of their group assignment because mechanical ventilation was initiated after anesthesia induction when they were unconscious. The anesthetic nurses and doctors evaluating the patients postoperatively were also unaware of the group assignments.

2.4. Anesthetic and analgesic managements Anesthesia was administered according to standardized institutional protocols. Patients received 1.5-2 mg/kg propofol, 1-2 mg/kg rocuronium, and 1-2 μg/kg remifentanil for induction. Anesthesia was maintained with inhaled sevoflurane or desflurane, with the inhaled concentration adjusted based on the electroencephalogram (EEG). Remifentanil was continuously infused at 0.05-0.2 μg/kg/min, adjusting blood pressure and heart rate to within ±20% of baseline values.

Thirty minutes before anesthesia emergence, all patients were administered 30 mg ketorolac tromethamine (Chengdu Dominant Pharmaceuticals Co., Ltd., China), 1 μg/kg fentanyl, and 4 mg tramadol (Jiangsu Hengrui Pharmaceuticals Co., Ltd., China), and a patient-controlled analgesia (PCA) device (Y-G-B3, JIANGSU YaGuang Medical Appliance CO., LTD., China) was initiated. The PCA was set to deliver a bolus dose of 15 μg fentanyl with a 10-minute lockout interval and no basal infusion (1 mg fentanyl and 8 mg tramadol mixed in 100 mL of normal saline solution). Data on PCA usage were collected, including the time and dose of each administration.

If the pain remained intolerable despite these measures, rescue analgesia was administered, including 1 μg/kg fentanyl or 30 mg ketorolac tromethamine IV.

2.5. Interventions Patients in the PCV group underwent mechanical ventilation in PC mode after induction. The ventilator (MAQUET Flow-I, MAQUET Italia S.p.A. Via Gozzano 14, 200 92 Cinisello Balsamo, (MI) Italy) settings were as follows: Adjust inspiratory pressure (Pins) to maintain the end-tidal carbon dioxide concentration (ETCO2) at 4.0-5.0 kPa. The investigators used 0.3 L/min of pure oxygen and air each, with an oxygen concentration of 41%.

Patients in the VCV group underwent mechanical ventilation in VC mode after induction. The ventilator was set with a tidal volume of 6-8 ml/kg, positive end-expiratory pressure (PEEP) at 0 cmH2O, a ratio of inspiration to expiration of 1:2, a respiratory rate of 16 breaths per minute, and an oxygen concentration of 41%.

Patients in the PRVC group underwent mechanical ventilation in PRVC mode after induction. The respiratory parameters were the same as those in group Ⅱ.

2.6. Outcome measures Record the following parameters at five time points: before insufflation (T1), 5 minutes after insufflation (T2), 10 minutes after insufflation (T3), 15 minutes after insufflation (T4), and 20 minutes after insufflation (T5). Esophageal pressure (pleural pressure, PES), mean airway pressure (PAWM), peak airway pressure (PAP), arterial carbon dioxide partial pressure (PaCO2), end-tidal carbon dioxide concentration (ETCO2), tidal volume (TV), mean arterial pressure (MAP; calculated as diastolic pressure + 1/3 pulse pressure), heart rate (HR), and optic nerve sheath diameter (ONSD). Since SpO2 was 100% at all time points for each group with no statistical difference, SpO2 is not included in the table.

Esophageal pressure (PES) was monitored using a Swan-Ganz catheter (Swan-Ganz, Edwards Lifesciences LLC, One Edwrds Way, Irvine, CA USA 92614) connected to a monitor (M8003A, Hewlett-Packard-Str. 2, 71034 Boblingen, Germany). Blood chemistry parameters were monitored using a blood gas analyzer (i-STAT1 Analyzer MN:300-G, Abbott Park, IL 60064 USA). Optic nerve sheath diameter (ONSD) was measured using an ultrasound system (On-platform ultrasound system PX, Vianen, Netherlands).

In the Postanesthetic Care Unit (PACU), record the following: Length of stay in PACU, Mean arterial pressure, Heart rate, Postoperative nausea and vomiting, Pain, Rescue antiemetics, Rescue analgesics, Rescue Sulfentanil dose.

2.7. Sample size The hypothesis of this study is that optic nerve sheath diameter (ONSD) can effectively differentiate between groups of different ventilation modes, with the hypothesis that the area under the ROC curve for ONSD is greater than 0.5. Preliminary experiments showed that the area under the ROC curve for ONSD is 0.7. With α=0.05 (one-tailed), β=0.1, and an equal ratio of 1:1:1 between groups, the sample size was estimated using n=Δ2/σ2(zα/2+zβ)2 [11,12]. It was found that at least 25 patients were needed per group. Considering a 20% dropout rate, the study included 30 patients in the PCV group, 30 in the VCV group, and 30 in the PRVC group.

2.8. Statistical analysis The sample size was estimated using the "Diagnostic Test (ROC)" - "Test for One Sample Sensitivity and Specificity" module in PASS 11 software. Data are presented as mean (standard deviation), frequency (%), or median (interquartile range). All statistical analyses were performed using GraphPad Prism version 10.2.3.The Kolmogorov-Smirnov test was performed to investigate the normality of the distribution of continuous variables. An independent t test or Mann-Whitney U test was performed to compare continuous variables, as appropriate. The x2 test or Fisher's exact was performed to compare categorical variables. Repeated-measures analysis of variance was performed to compare changes in some variables over time. Statistical significance was set at P value <0.05.

ELIGIBILITY:
Inclusion Criteria:

●The patients had an ASA classification of I-III.

Exclusion Criteria:

* allergy to the anesthetic drugs
* liver cirrhosis
* kidney dysfunction
* cardiopulmonary impairment
* Patients were uncooperative

Ages: 22 Years to 77 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study enrolled patients who underwent elective laparoscopic myomectomy.
Enrollment: 90 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Average Airway Pressure (PAWM) in the Trendelenburg Position | Measurements will be taken at five specific time points: before and after pneumoperitoneum at 5, 10, 15, and 20 minutes.
  The normal range for Average Airway Pressure (PAWM) during mechanical ventilation is 5-10 cmH2O. The higher the value, the greater the pressure, and the worse the outcome.
Optic Nerve Sheath Diameter (ONSD) as a Measure of Intracranial Pressure | ONSD measurements will be recorded at the same five time points as PAWM: before and after pneumoperitoneum at 5, 10, 15, and 20 minutes.
  Optic Nerve Sheath Diameter (ONSD) is a non-invasive method used to assess increased intracranial pressure through ultrasonographic measurement. The normal range for ONSD is approximately between 3.3mm and 5.2mm, while a value exceeding 5mm is generally considered indicative of possible increased intracranial pressure.

SECONDARY OUTCOMES:
Hemodynamic Stability as Assessed by Mean Arterial Pressure (MAP) and Heart Rate (HR) | MAP and HR will be recorded at the same five time points as PAWM and ONSD: before and after pneumoperitoneum at 5, 10, 15, and 20 minutes.
  Mean Arterial Pressure (MAP), the normal MAP value for adults is typically between 70 to 105mmHg. A MAP exceeding 105 indicates light anesthesia, while below 70 suggests deep anesthesia. Heart Rate (HR), the standard heart rate range for adults at rest is usually 60 to 100 beats per minute. An HR exceeding 100 indicates light anesthesia, and below 60 suggests deep anesthesia. Deviations of MAP and HR from the normal range are undesirable outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
Esophageal pressure (pleural pressure, PES), mean airway pressure (PAWM), peak airway pressure (PAP), arterial carbon dioxide partial pressure (PaCO2), end-tidal carbon dioxide concentration (ETCO2), tidal volume (TV), mean arterial pressure (MAP; calculated as diastolic pressure + 1/3 pulse pressure), heart rate (HR), and optic nerve sheath diameter (ONSD).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: from February 2023 to August 2033
Access Criteria: Anyone